CLINICAL TRIAL: NCT06257992
Title: Effectiveness of Dry Needling of Active Trigger Points in Neck Muscles in Patients With Chronic Cervical Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Julian Müller-Thyssen Uriarte, Principal Investigator, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RAT 2022-53
Record Dates: First submitted 2024-02-05; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Cervical Pain
MeSH Terms: conditions — Neck Pain | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling Group (Experimental)
  Interventions: Other: Dry Needling
- Stretch Group (Active Comparator)
  Interventions: Other: Stretch

INTERVENTIONS:
Other: Dry Needling — 3 treatments of dry needling to inactivate all active trigger points found in patient's cervical muscles.
  Arms: Dry Needling Group
Other: Stretch — 3 treatments of stretch applied to all cervical muscles that present active trigger points in patient's cervical muscles.
  Arms: Stretch Group

SUMMARY:
Randomized Single-Blind Clinical Trial in which the treatment will be administered through 3 sessions of dry needling in the cervical muscles's active trigger points in patients with chronic cervical pain.

ELIGIBILITY:
Inclusion Criteria:

* Be older than 18 years old
* Sign informed consent form prior to participating in this study
* Have chronic cervical pain diagnosis of their primary care doctor.
* Have one or more active myofascial trigger point in the cervical muscles according to the criteria established by Simons et al.

Exclusion Criteria:

* Major trauma on cervical spine stated from the medical history
* Inflammatory, hormonal or neurological disorders
* Have contraindication to conservative or invasive physiotherapy (infection, fever, hypothyroidism, wound in the puncture area, metal allergies, cancer or systemic diseases, or belonephobia)
* Having received physiotherapy treatment for the condition in the past month

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Cervical Pain Intensity | Change between baseline (immediately before intervention) and post intervention (immediately after intervention), after 1month and 3 months
  For the Assesment of cervical pain intensity the Numeric Pain Rating Scale (NPRS) was used.
Neck Disability Index | Change between baseline (immediately before intervention) and post intervention (immediately after intervention), after 1month and 3 months
  For the assesment of perceived neck disability the neck disability index was used.
Pressure Pain Threshold | Change between baseline (immediately before intervention) and post intervention (immediately after intervention), after 1month and 3 months
  For the assesment of pressure pain threshold of active trigger points a digital algometer was used

SECONDARY OUTCOMES:
Cervical range of movement | Change between baseline (immediately before intervention) and post intervention (immediately after intervention), after 1month and 3 months
  For the assesment of cervical range of movement the universal goniometer was used
Cervical muscles Electromyography | Change between baseline (immediately before intervention) and post intervention (immediately after intervention), after 1month and 3 months
  For the assesment of cervical muscles electromyographic activity Trigno Avanti sensor was used.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Clínico de Fisioterapia OMT-E, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cerezo-Tellez E, Torres-Lacomba M, Fuentes-Gallardo I, Perez-Munoz M, Mayoral-Del-Moral O, Lluch-Girbes E, Prieto-Valiente L, Falla D. Effectiveness of dry needling for chronic nonspecific neck pain: a randomized, single-blinded, clinical trial. Pain. 2016 Sep;157(9):1905-1917. doi: 10.1097/j.pain.0000000000000591. PMID 27537209
- [Background] Fernandez-de-las-Penas C, Alonso-Blanco C, Miangolarra JC. Myofascial trigger points in subjects presenting with mechanical neck pain: a blinded, controlled study. Man Ther. 2007 Feb;12(1):29-33. doi: 10.1016/j.math.2006.02.002. PMID 21882489
- [Background] Navarro-Santana MJ, Sanchez-Infante J, Gomez-Chiguano GF, Cleland JA, Fernandez-de-Las-Penas C, Martin-Casas P, Plaza-Manzano G. Dry Needling Versus Trigger Point Injection for Neck Pain Symptoms Associated with Myofascial Trigger Points: A Systematic Review and Meta-Analysis. Pain Med. 2022 Mar 2;23(3):515-525. doi: 10.1093/pm/pnab188. PMID 34114639
- [Background] Ball AM, Finnegan M, Koppenhaver S, Freres W, Dommerholt J, Mayoral Del Moral O, Bron C, Moore R, Ball EE, Gaffney EE. The relative risk to the femoral nerve as a function of patient positioning: potential implications for trigger point dry needling of the iliacus muscle. J Man Manip Ther. 2019 Jul;27(3):162-171. doi: 10.1080/10669817.2019.1568699. Epub 2019 Feb 20. PMID 30935326